CLINICAL TRIAL: NCT02448589
Title: A Phase I, Open-Label, Non-Randomized, Dose-Escalating Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of TAS-119 in Patients With Advanced Solid Tumors
Brief Title: An Investigation of TAS-119 Monotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-119-102; 2014-001272-63 (EudraCT Number)
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Dose Escalation; Dose Expansion; MTD; TAS-119; Aurora A Kinase Inhibitor
MeSH Terms: interventions — TAS-119

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAS-119 Monotherapy (Experimental): Dose Escalation:
  A Monotherapy Dose-Escalation Phase Performed in Approximately 5 Dose Levels (3 to 12 Patients Per Dose Level) to Determine the MTD for TAS-119 Given Orally (PO), Twice-Daily (BID) in a 28-Day Treatment Cycle; and:
  Dose Expansion:
  A Monotherapy Expansion Phase in Which Approximately 40 Additional Patients will be Enrolled to Further Evaluate the Recommended Phase II Dose (RP2D)
  Interventions: Drug: TAS-119

INTERVENTIONS:
Drug: TAS-119

SUMMARY:
A Phase 1, Open-Label, Non-Randomized, Dose-Escalating Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of TAS-119 in Patients with Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, dose escalation study of TAS-119 evaluating the safety, tolerability, PK, pharmacogenomics, pharmacodynamics, and preliminary antitumour activity in patients with advanced and unresectable solid tumours. The study will evaluate TAS-119 monotherapy, employing two sequential phases.

* A Dose Escalation Phase
* An Expansion Phase

ELIGIBILITY:
Inclusion criteria include the following:

1. Is a male or female, ≥ 18 years of age, who has provided written informed consent.
2. Has histologically or cytologically confirmed advanced, unresectable, metastatic solid tumor(s) for which the patients have no available therapy likely to provide clinical benefit.
3. Must have an archival FFPE tumor sample available, to be provided to the Sponsor upon request.
4. In the Expansion Phase: patients should be willing to undergo tumor core biopsy procedure at pre-treatment and on Day 4, Cycle 1 if, in the judgment of the investigator, it is considered clinically safe and appropriate to do so. This requirement is optional but preferred for patients in Dose Escalation.
5. Has adequate organ function.

Women of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug. Both males and females and must agree to use effective birth control during the study if conception is possible during this interval.

Exclusion:

1. Has received prior treatment with TAS-119.
2. Has received treatment with any proscribed treatments within specified time frames prior to study drug administration.
3. Has a serious illness or medical condition(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Up to 2.5 Years
  Identify the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of TAS-119

CONTACTS AND LOCATIONS:
Locations (6):
- University Hospitals - Seidman Cancer Center, Cleveland, Ohio, United States
- San Raffaele Hospital, Milan, Italy
- Erasmus MC Cancer Institute, Rotterdam, Netherlands
- Spain (2):
  - START MADRID-FJD, Hospital Fundación Jiménez Díaz, Madrid
  - START Madrid Unidad de Ensayos Fase I, Madrid
- The Institute of Cancer Research, Sutton, Surrey, United Kingdom

REFERENCES:
- [Background] Mountzios G, Terpos E, Dimopoulos MA. Aurora kinases as targets for cancer therapy. Cancer Treat Rev. 2008 Apr;34(2):175-82. doi: 10.1016/j.ctrv.2007.09.005. Epub 2007 Nov 19. PMID 18023292
- [Background] Ogawa E, Takenaka K, Katakura H, Adachi M, Otake Y, Toda Y, Kotani H, Manabe T, Wada H, Tanaka F. Perimembrane Aurora-A expression is a significant prognostic factor in correlation with proliferative activity in non-small-cell lung cancer (NSCLC). Ann Surg Oncol. 2008 Feb;15(2):547-54. doi: 10.1245/s10434-007-9653-8. Epub 2007 Nov 28. PMID 18043979
- [Background] Xu HT, Ma L, Qi FJ, Liu Y, Yu JH, Dai SD, Zhu JJ, Wang EH. Expression of serine threonine kinase 15 is associated with poor differentiation in lung squamous cell carcinoma and adenocarcinoma. Pathol Int. 2006 Jul;56(7):375-80. doi: 10.1111/j.1440-1827.2006.01974.x. PMID 16792546
- [Background] Nadler Y, Camp RL, Schwartz C, Rimm DL, Kluger HM, Kluger Y. Expression of Aurora A (but not Aurora B) is predictive of survival in breast cancer. Clin Cancer Res. 2008 Jul 15;14(14):4455-62. doi: 10.1158/1078-0432.CCR-07-5268. PMID 18628459
- [Background] Lassmann S, Shen Y, Jutting U, Wiehle P, Walch A, Gitsch G, Hasenburg A, Werner M. Predictive value of Aurora-A/STK15 expression for late stage epithelial ovarian cancer patients treated by adjuvant chemotherapy. Clin Cancer Res. 2007 Jul 15;13(14):4083-91. doi: 10.1158/1078-0432.CCR-06-2775. PMID 17634533
- [Background] Lagarde P, Perot G, Kauffmann A, Brulard C, Dapremont V, Hostein I, Neuville A, Wozniak A, Sciot R, Schoffski P, Aurias A, Coindre JM, Debiec-Rychter M, Chibon F. Mitotic checkpoints and chromosome instability are strong predictors of clinical outcome in gastrointestinal stromal tumors. Clin Cancer Res. 2012 Feb 1;18(3):826-38. doi: 10.1158/1078-0432.CCR-11-1610. Epub 2011 Dec 13. PMID 22167411
- [Background] Reiter R, Gais P, Jutting U, Steuer-Vogt MK, Pickhard A, Bink K, Rauser S, Lassmann S, Hofler H, Werner M, Walch A. Aurora kinase A messenger RNA overexpression is correlated with tumor progression and shortened survival in head and neck squamous cell carcinoma. Clin Cancer Res. 2006 Sep 1;12(17):5136-41. doi: 10.1158/1078-0432.CCR-05-1650. PMID 16951231
- [Background] Anand S, Penrhyn-Lowe S, Venkitaraman AR. AURORA-A amplification overrides the mitotic spindle assembly checkpoint, inducing resistance to Taxol. Cancer Cell. 2003 Jan;3(1):51-62. doi: 10.1016/s1535-6108(02)00235-0. PMID 12559175
- [Background] McGrogan BT, Gilmartin B, Carney DN, McCann A. Taxanes, microtubules and chemoresistant breast cancer. Biochim Biophys Acta. 2008 Apr;1785(2):96-132. doi: 10.1016/j.bbcan.2007.10.004. Epub 2007 Nov 12. PMID 18068131
- [Background] Beltran H, Rickman DS, Park K, Chae SS, Sboner A, MacDonald TY, Wang Y, Sheikh KL, Terry S, Tagawa ST, Dhir R, Nelson JB, de la Taille A, Allory Y, Gerstein MB, Perner S, Pienta KJ, Chinnaiyan AM, Wang Y, Collins CC, Gleave ME, Demichelis F, Nanus DM, Rubin MA. Molecular characterization of neuroendocrine prostate cancer and identification of new drug targets. Cancer Discov. 2011 Nov;1(6):487-95. doi: 10.1158/2159-8290.CD-11-0130. PMID 22389870
- [Background] Tajiri T, Tanaka S, Shono K, Kinoshita Y, Fujii Y, Suita S, Ihara K, Hara T. Quick quantitative analysis of gene dosages associated with prognosis in neuroblastoma. Cancer Lett. 2001 May 10;166(1):89-94. doi: 10.1016/s0304-3835(01)00434-7. PMID 11295291
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Brockmann M, Poon E, Berry T, Carstensen A, Deubzer HE, Rycak L, Jamin Y, Thway K, Robinson SP, Roels F, Witt O, Fischer M, Chesler L, Eilers M. Small molecule inhibitors of aurora-a induce proteasomal degradation of N-myc in childhood neuroblastoma. Cancer Cell. 2013 Jul 8;24(1):75-89. doi: 10.1016/j.ccr.2013.05.005. Epub 2013 Jun 20. PMID 23792191
- [Background] Kalliokoski A, Niemi M. Impact of OATP transporters on pharmacokinetics. Br J Pharmacol. 2009 Oct;158(3):693-705. doi: 10.1111/j.1476-5381.2009.00430.x. Epub 2009 Sep 25. PMID 19785645
- [Background] Niemi M, Pasanen MK, Neuvonen PJ. Organic anion transporting polypeptide 1B1: a genetically polymorphic transporter of major importance for hepatic drug uptake. Pharmacol Rev. 2011 Mar;63(1):157-81. doi: 10.1124/pr.110.002857. Epub 2011 Jan 18. PMID 21245207
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Bogaerts J, Ford R, Sargent D, Schwartz LH, Rubinstein L, Lacombe D, Eisenhauer E, Verweij J, Therasse P; RECIST Working Party. Individual patient data analysis to assess modifications to the RECIST criteria. Eur J Cancer. 2009 Jan;45(2):248-60. doi: 10.1016/j.ejca.2008.10.027. Epub 2008 Dec 16. PMID 19095437
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Raphael C, Briscoe C, Davies J, Ian Whinnett Z, Manisty C, Sutton R, Mayet J, Francis DP. Limitations of the New York Heart Association functional classification system and self-reported walking distances in chronic heart failure. Heart. 2007 Apr;93(4):476-82. doi: 10.1136/hrt.2006.089656. Epub 2006 Sep 27. PMID 17005715
- [Derived] Robbrecht DGJ, Lopez J, Calvo E, He X, Hiroshi H, Soni N, Cook N, Dowlati A, Fasolo A, Moreno V, Eskens FALM, de Bono JS. A first-in-human phase 1 and pharmacological study of TAS-119, a novel selective Aurora A kinase inhibitor in patients with advanced solid tumours. Br J Cancer. 2021 Jan;124(2):391-398. doi: 10.1038/s41416-020-01100-3. Epub 2020 Oct 6. PMID 33020594